CLINICAL TRIAL: NCT06331858
Title: The Effect of Adding Instrumented Hip Concentric Abductor Strengthening Exercise to Instrumented Knee Flexor-Extensor Concentric Strengthening Exercise on Pain, Function, Physical Performance, and Quality of Life in Knee Osteoarthritis
Brief Title: The Effect of Adding Instrumented Hip Concentric Abductor Strengthening Exercise in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Hasan Hüseyin Gökpınar, Assistant professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KutahyaHSU-DRGOKPINARDROMER-43
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis; Pain; Physical Disability
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: 1. STUDY GROUP
  2. CONTROL GROUP
Who Masked: Investigator, Outcomes Assessor
Masking Description: Before and after the treatment, all patients were evaluated by a blind evaluator in terms of physical examination, pain and functionality, physical performance, quality of life and gait parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Active Comparator): The study group received hip device-assisted concentric abductor strengthening (HDACAS) program in addition to knee device-assisted concentric flexor-extensor strengthening (KDACFES) program.
  Interventions: Device: hip device-assisted concentric abductor strengthening (HDACAS); Device: knee device-assisted concentric flexor-extensor strengthening (KDACFES)
- Control group (Active Comparator): The control group received only KDACFES program
  Interventions: Device: knee device-assisted concentric flexor-extensor strengthening (KDACFES)

INTERVENTIONS:
Device: hip device-assisted concentric abductor strengthening (HDACAS) — All participants received device-assisted strengthening exercises with increasing doses according to a pre-determined strengthening program for a total of 6 weeks, 4 days a week, and a total of 24 sessions
  Arms: Study group
Device: knee device-assisted concentric flexor-extensor strengthening (KDACFES) — All participants received device-assisted strengthening exercises with increasing doses according to a pre-determined strengthening program for a total of 6 weeks, 4 days a week, and a total of 24 sessions

SUMMARY:
The aim of this study was to investigate the effectiveness of adding hip device-assisted concentric abductor strengthening (HDACAS) program to knee device-assisted concentric flexor-extensor strengthening (KDACFES) program on pain, function, physical performance, quality of life and gait parameters in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This prospective randomized single-blind controlled study was conducted at Kütahya Health Sciences University (KHSU) Evliya Çelebi Education and Research Hospital (ECERH) Physical Medicine and Rehabilitation (PMR) annex building between September 2023 and March 2024. The study protocol was approved by the ethics committee of the same university (2023-03/03).

ELIGIBILITY:
Inclusion Criteria:

* Receiving a diagnosis of knee osteoarthritis according to the ACR criteria and being classified as stage 2-3 according to the Kellgren Lawrence staging
* Having symptomatic unilateral or bilateral knee pain with a VAS (0-10) pain score > 4
* Being able to ambulate independently without orthosis/prosthesis
* Having a body mass index less than 35

Exclusion Criteria:

* History of knee and hip surgery
* Presence of lesions, atrophy, or scars in the skin area
* Intra-articular injection to the knee within the last 6 months
* Receiving active physiotherapy, physical therapy, or spa treatment in the last 6 months
* Patients with chronic diseases such as COPD, coronary artery disease
* Those with oxygen saturation levels <95%
* Individuals with any pathological condition that may impair normal walking
* Patients with diseases such as vertigo, epilepsy that may pose a risk during physical performance tests
* Patients with contraindications to strength training exercises

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities (WOMAC) | TIME FRAME 1: pre-intervention (up to 72 hours), TIME FRAME 2: post-intervention(up to 72 hours)
  Assessments consist of three components: pain, stiffness, and functionality. The WOMAC consists of three subscales: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Scores range from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status. The higher the score, the poorer the function.
The Lequesne Algofunctional index | TIME FRAME 1: pre-intervention (up to 72 hours), TIME FRAME 2: post-intervention(up to 72 hours)
  It is a disease-specific measure used to assess the pain, maximum walking distance, and daily life activities of knee osteoarthritis patients.
  The Lequesne Algofunctional index has an interview format questionnaire, including 10 questions divided into three sections regarding pain, maximum distance walked and activities of daily living. The score ranges from 0 (no pain, no disability) to 24 (maximum pain and disability.
TIME UP AND GO TEST | TIME FRAME 1: pre-intervention (up to 72 hours), TIME FRAME 2: post-intervention(up to 72 hours)
  With this test, patients' ability to maintain balance during transfer and walking is assessed. One source suggests that scores of ten seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention.
30 SECOND CHAIR TEST | TIME FRAME 1: pre-intervention (up to 72 hours), TIME FRAME 2: post-intervention(up to 72 hours)
  This test requires the individual to sit and stand continuously for 30 seconds with arms crossed over the chest and is based on the maximum number of repetitions the individual can perform. The 30-second chair stand involves recording the number of stands a person can complete in 30 seconds rather then the amount of time it takes to complete a pre-determined number of repetitions.Great: 19 or more reps in 30 seconds means your endurance and lower-body strength are above average. You have the greatest life expectancy. Average: Between 10 and 18 reps indicates average endurance and lower-body strength. Poor: 9 reps or fewer should be considered a warning sign.
40 METER SELF PACED WALK TEST | TIME FRAME 1: pre-intervention (up to 72 hours), TIME FRAME 2: post-intervention(up to 72 hours)
  It is a test focused on measuring mobility and function. It is based on walking a certain distance in the fastest possible time, competing against time. A fast-paced walking test that is timed over 4 x 10m (33 ft) for a total 40 m (132 ft) (2). As a direct measure of the ability to walk quickly over short distances, which is an activity that is important but often limited in people with hip and/or knee OA. Regular walking aid is allowed and recorded. Time of one trial, with turn time excluded, is recorded and expressed as speed m/s by dividing distance (40 m) by time (s)
SIX MINUTES WALK TEST | TIME FRAME 1: pre-intervention (up to 72 hours), TIME FRAME 2: post-intervention(up to 72 hours)
  The 6-minute walk test, which is a reliable and valid mobility test for measuring walking activity, is the most commonly used test in clinical trials. The maximum distance that can be walked over a 6-min interval is recorded. Rest periods are allowed but included in the time Standardized encouragement (e.g., keep going you are doing really well") can be given at minute intervals. Regular walking aid is allowed. Practice test not needed in most clinical settings but if performed then at least 1 h rest should be allowed before the second test. The greatest distance is then recorded
STAIR CLIMB TEST | TIME FRAME 1: pre-intervention (up to 72 hours), TIME FRAME 2: post-intervention(up to 72 hours)
  It is a test that varies in the number of steps, but the most commonly used and the version found on the OARSI website is the 9-step stair climb test. Ascend and descend flight of nine stairs in a usual manner, and at a safe and comfortable pace. Use of any walking aid and handrail is permitted and recorded. Total time to ascend and descend steps for one trial is recorded in seconds

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | TIME FRAME 1: pre-intervention (up to 72 hours), TIME FRAME 2: post-intervention(up to 72 hours)
  The intensity of pain ranges from '0' to '10', with '0' indicating no pain and '10' representing the worst pain the person has ever experienced in their life
Mini Osteoarthritis Knee and Hip Quality of Life Scale | TIME FRAME 1: pre-intervention (up to 72 hours), TIME FRAME 2: post-intervention(up to 72 hours)
  It is derived from the original Osteoarthritis Knee and Hip Quality of Life (OAKHQoL) questionnaire, developed to assess Health-Related Quality of Life (HRQoL) in patients with knee and/or hip osteoarthritis. It includes five subscales: physical activities, mental health, pain, social support, social functioning; with three additional independent items addressing sexual life, professional life, and fear of being dependent. The numerical rating scales in the items range from 0 (worst) to 10 (best). Scores were obtained by computing the means of the item scores in each subscale. The last three items' score (independent items) becomes the corresponding score.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan H Gökpınar, Study Director — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Kütahya, Turkey (Türkiye)